CLINICAL TRIAL: NCT03061266
Title: The Application of the E-health Education on Shared Care Program for Patients With Type 2 Diabetes - Taking Local Teaching Hospital for Example
Brief Title: The Application of the E-health Education on Shared Care Program for Patients With Type 2 Diabetes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Li-Li Chen (Other)
Responsible Party: Sponsor-Investigator, Li-Li Chen, Principal Investigator, China Medical University Hospital
Organization: China Medical University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: CMUH105-REC2-013
Record Dates: First submitted 2017-02-19; First posted 2017-02-23 (Actual); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: type 2 diabetes mellitus, application, e-health education
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- E-health education group (Experimental): E-health education group will be received the shared care program using e-health education.
  Interventions: Behavioral: E-health Education
- Routine care (Other): Control group will be received the shared care program as advised by clinical professionals, which included medications, dietary control and general physical activities.
  Interventions: Other: Routine care

INTERVENTIONS:
Behavioral: E-health Education — E-health education on shared care program will be established by different type's professionals including diabetes physicians, pharmacists, dietitians and diabetes health teacher.
  Arms: E-health education group
Other: Routine care — Routine care on shared care program as advised by clinical professionals, which included medications, dietary control and general physical activities.
  Arms: Routine care

SUMMARY:
This study will be a randomized controlled trial aimed at examining the effectiveness of the in e-health education on shared care program for patients with type 2 diabetes mellitus (T2DM). The experiment will be conducted over 1 year at a regional hospital in Taiwan. The research subjects will be excluded 160 patients with T2DM. Subjects assigned to an experimental group will receive the integrated care program, whereas those assigned to a control group will receive routine care. The membership of e-health education on shared care program is established by different type's professionals including diabetes physicians, pharmacists, dietitians and diabetes health teacher. Glycated hemoglobin (HbA1c) of subjects in both groups will be measured at three time points including 1 month before the experiment, and 2 and 5 months after the experiment. The self-management conditions and quality of life of the subjects will be also recorded using relevant scales.

DETAILED DESCRIPTION:
This study will be a randomized controlled trial aimed at examining the effectiveness of the in e-health education on shared care program for patients with type 2 diabetes mellitus (T2DM). The experiment will be conducted over 1 year at a regional hospital in Taiwan. The research subjects will be excluded 160 patients with T2DM. Subjects assigned to an experimental group will receive the integrated care program, whereas those assigned to a control group will receive routine care. The membership of e-health education on shared care program is established by different type's professionals including diabetes physicians, pharmacists, dietitians and diabetes health teacher. Glycated hemoglobin (HbA1c) of subjects in both groups will be measured at three time points including 1 month before the experiment, and 2 and 5 months after the experiment. The self-management conditions and quality of life of the subjects will be also recorded using relevant scales. SPSS+ 22.0 statistics software will be used for a statistical analysis, which will be presented in percentages, means, and standard deviations. Additionally, the chi-square test will be also to examine the homogeneity of both groups. Generalized estimating equations will be used to analyze repeated measurements in order to compare the efficacy of improving HbA1c, self-management, and quality of life. We anticipate that the results of this study will provide the e-health education on shared care program to clinical nursing staff to assist patients with T2DM in controlling their blood sugar as well as to improve their self-management and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* participation with type 2 diabetes mellitus received oral medication.

Exclusion Criteria:

* Studies were excluded from this study if participation had recently undergone serious operations, had a myocardial infarction, stroke, severe liver or kidney diseases, received injection medication,or any illness limiting participation in a physical activity program.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2016-03-09 (Actual); Primary Completion 2017-03-08 (Estimated); Study Completion 2017-03-08 (Estimated)

PRIMARY OUTCOMES:
Glycated hemoglobin (HbA1c) | up to 6 months after the experiment
  glucose index

SECONDARY OUTCOMES:
Perceived diabetes self-management abilty using questionnaire | baseline, 3 and 6 months after the experiment
  self-management abilty
quality of life using questionnaire | baseline, 3 and 6 months after the experiment
  the general well-being of individuals and societies, outlining negative and positive features of life

CONTACTS AND LOCATIONS:
Overall Officials: Chen Li-Li, PhD, Study Director — China Medical University, Taichung, Taiwan; Pai Lee-Wen, PhD, Principal Investigator — Department of Nursing, Central Taiwan University of Science and Technology, Taichung, Taiwan
Locations (1):
- Puli Christian Hospital, Nantou City, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Frederick V, Matilda SA, Margaret AK, Seth A. Population-based study of diabetic mellitus prevalence and its associated factors in adult Ghanaians in the greater Accra region. International Journal of Diabetes in Developing Countries. 2011; 31:149-53.
- [Background] Lin CC, Li CI, Hsiao CY, Liu CS, Yang SY, Lee CC, Li TC. Time trend analysis of the prevalence and incidence of diagnosed type 2 diabetes among adults in Taiwan from 2000 to 2007: a population-based study. BMC Public Health. 2013 Apr 9;13:318. doi: 10.1186/1471-2458-13-318. PMID 23570503
- [Background] Shen FC, Chen CY, Su SC, Liu RT. The Prevalence and Risk Factors of Diabetic Nephropathy in Taiwanese Type 2 Diabetes-A Hospital-Based Study. Acta Nephrologica. 2009; 23:90-95.
- [Background] World Health Organization. National Diabetes Fact Sheet 2015. 2015. Available at http://www.who.int/mediacentre/factsheets/fs312/en/index.html. Last accessed 4 May 2015.
- [Result] American Diabetes Association. Standards of medical care in diabetes--2013. Diabetes Care. 2013 Jan;36 Suppl 1(Suppl 1):S11-66. doi: 10.2337/dc13-S011. No abstract available. PMID 23264422
- [Result] Beard E, Clark M, Hurel S, Cooke D. Do people with diabetes understand their clinical marker of long-term glycemic control (HbA1c levels) and does this predict diabetes self-care behaviours and HbA1c? Patient Educ Couns. 2010 Aug;80(2):227-32. doi: 10.1016/j.pec.2009.11.008. Epub 2009 Dec 24. PMID 20036098
- [Result] Bhatti S A, Khan A H, Yaqoob N. Glycated hemoglobin(HbA1c);screening for undiagnosed diasetes in healthy individuals in Sargodha. The Professional Medical Journal.2015; 22(2):208-214.
- [Result] Cheung NW, Yue DK, Kotowicz MA, Jones PA, Flack JR. A comparison of diabetes clinics with different emphasis on routine care, complications assessment and shared care. Diabet Med. 2008 Aug;25(8):974-8. doi: 10.1111/j.1464-5491.2008.02522.x. PMID 18959612
- [Result] Breen GM, Zhang NJ. Introducing ehealth to nursing homes: theoretical analysis of improving resident care. J Med Syst. 2008 Apr;32(2):187-92. doi: 10.1007/s10916-007-9121-9. PMID 18461822
- [Result] Chiou ST, Lin HD, Yu NC, Hseuh HK, Lin LH, Lin LT, Chen TJ, Lai MS. An initial assessment of the feasibility and effectiveness of implementing diabetes shared care system in Taiwan--some experiences from I-Lan County. Diabetes Res Clin Pract. 2001 Nov;54 Suppl 1:S67-73. doi: 10.1016/s0168-8227(01)00311-4. PMID 11580971
- [Result] Graffigna G, Barello S, Bonanomi A, Menichetti J. The Motivating Function of Healthcare Professional in eHealth and mHealth Interventions for Type 2 Diabetes Patients and the Mediating Role of Patient Engagement. J Diabetes Res. 2016;2016:2974521. doi: 10.1155/2016/2974521. Epub 2016 Jan 5. PMID 26881243
- [Result] Pacaud D., Kelley H, Downey A , Chiasson M. Successful Delivery of Diabetes Self-Care Education and Follow-Up through eHealth Media. Canadian Journal of Diabetes 2012; 36(5): 257-262.
- [Result] Sacks DB, Arnold M, Bakris GL, Bruns DE, Horvath AR, Kirkman MS, Lernmark A, Metzger BE, Nathan DM; National Academy of Clinical Biochemistry. Position statement executive summary: guidelines and recommendations for laboratory analysis in the diagnosis and management of diabetes mellitus. Diabetes Care. 2011 Jun;34(6):1419-23. doi: 10.2337/dc11-9997. PMID 21617111